CLINICAL TRIAL: NCT01971333
Title: The Validity of Dynamic Preload Parameters During Liver Transplantation
Brief Title: Dynamic Preload Parameters During Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201309024RIND
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Liver Cirrhosis
Keywords: pulse pressure variation; stroke volume variation; plethysmographic variation index; fluid responsiveness
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liver transplantation: Compare intraoperative change of dynamic parameters after fluid loading:
  1. pulse pressure variation
  2. stroke volume variation
  3. plethysmographic variation index

SUMMARY:
The arterial system compliance is compromised in liver cirrhotic patients. Dynamic preload variables are either pressure-based (e.g.pulse pressure variation; PPV), flow-based (e.g. stroke volume variation; SVV), or volume-based (plethysmographic variability index; PVI). It is not yet clear that dynamic preload parameters based on which mechanism will be accurate to predict fluid responsiveness in the cirrhotic patients. Therefore, this study aimed to claried which dynamic preload parameters would be more accurate during the liver transplantation.

DETAILED DESCRIPTION:
Fluid management is crucial during liver transplantation. Patients with cirrhosis and portal hypertension have an altered blood volume distribution and pooling in the splanchnic circulation. Excess administration of intravenous fluid may increase portal hypertension due to splanchnic venous congestion and may also aggravate coagulopathy by dilution. On the other hand, fluid restriction may risk systemic and especially renal hypoperfusion. Traditional static fluid parameter, such as central venous pressure, pulmonary artery occlusion pressure, have been reported inaccurate to predict fluid responsiveness. In comparison, the recent developed dynamic fluid parameters based on heart-lung interaction were reported to be good preload indicators in a variety of different surgical settings. However, the validity of such dynamic fluid parameters is highly dependent on The arterial system compliance is compromised in liver cirrhotic patients. Dynamic preload variables are either pressure-based (e.g.pulse pressure variation; PPV), flow-based (e.g. stroke volume variation; SVV), or volume-based (plethysmographic variability index; PVI). It is not yet clear that dynamic preload parameters based on which mechanism will be accurate to predict fluid responsiveness in the cirrhotic patients. Therefore, this study aimed to claried which dynamic preload parameters would be more accurate during the liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* End stage liver disease patients scheduled for liver transplantation in National Taiwan University Hospital

Exclusion Criteria:

* Allergic reaction
* preexisting arrythmia

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: End stage liver disease patients scheduled for liver transplantation in National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Change of cardiac index after fluid loading | one day

SECONDARY OUTCOMES:
Fluid responsiveness parameters: pulse pressure variation | one day
Fluid responsiveness parameters: stroke volume variation | one day
Fluid responsiveness parameters: plethysmographic variation index | one day

OTHER OUTCOMES:
Mean arterial pressure changes | one day
Central venous pressure changes | one day
Heart rate changes | one day

CONTACTS AND LOCATIONS:
Overall Officials: Chun Yu Wu, M.D., Principal Investigator — Department of Anesthesiology, National Taiwan University Hospital
Locations (1):
- Department of Anesthesiology, NTUH, Taipei, Taiwan, Taipei, Taiwan

REFERENCES:
- [Background] Vos JJ, Kalmar AF, Struys MM, Wietasch JK, Hendriks HG, Scheeren TW. Comparison of arterial pressure and plethysmographic waveform-based dynamic preload variables in assessing fluid responsiveness and dynamic arterial tone in patients undergoing major hepatic resection. Br J Anaesth. 2013 Jun;110(6):940-6. doi: 10.1093/bja/aes508. Epub 2013 Jan 24. PMID 23348202
- [Derived] Wu CY, Cheng YJ, Liu YJ, Wu TT, Chien CT, Chan KC; NTUH Center of Microcirculation Medical Research (NCMMR). Predicting stroke volume and arterial pressure fluid responsiveness in liver cirrhosis patients using dynamic preload variables: A prospective study of diagnostic accuracy. Eur J Anaesthesiol. 2016 Sep;33(9):645-52. doi: 10.1097/EJA.0000000000000479. PMID 27167058